CLINICAL TRIAL: NCT01948024
Title: An Open-label, Randomized, Two Treatment, Multi-site, Multiple Dose, Steady State, Three-way, Reference-replicated Crossover, Pharmacokinetic Study to Determine the In-vivo Bioequivalence Between Asenapine 10 mg Sublingual Tablet and SAPHRIS® (Asenapine) 10 mg Sublingual Tablet
Brief Title: Bio-equivalence Study Between SAPHRIS and Asenapine
Acronym: ASN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASN-101
Record Dates: First submitted 2013-08-09; First posted 2013-09-23 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference Arm - SAPHRIS (Active Comparator): 10 mg BID sublingual tablet
  Interventions: Drug: SAPHRIS
- Test Arm - Asenapine (Experimental): 10 mg BID sublingual tablet
  Interventions: Drug: Asenapine

INTERVENTIONS:
Drug: SAPHRIS — 10 mg BID sublingual tablet
  Arms: Reference Arm - SAPHRIS
Drug: Asenapine — 10 mg BID sublingual tablet
  Arms: Test Arm - Asenapine

SUMMARY:
This is a Multiple-dose, steady state, three-way reference-replicated crossover study.

The purpose of this Study is to determine the bio-equivalence between SAPHRIS and Asenapine 10mg sublingual tablets.

DETAILED DESCRIPTION:
Molecule Name Asenapine Country of submission US

PRODUCT DETAILS

Test formulation

Drug name: Asenapine Sublingual Tablet EQ 10mg base Manufactured by: Sun Pharmaceutical Industries, Ltd.

Reference formulation

Drug name: SAPHRIS® (Asenapine) sublingual tablets Manufactured by: Schering Corporation, a Subsidiary of Merck & Co., Inc.

STUDY DESIGN

Title An open-label, randomized, two treatment, multi-site, multiple dose, steady state, three-way, reference-replicated crossover, pharmacokinetic study to determine the in-vivo bioequivalence between Asenapine 10 mg sublingual tablet and SAPHRIS® (asenapine) 10 mg sublingual tablet

Study Design Multiple-dose, steady state, three-way reference-replicated crossover study

Type of Study Pharmacokinetic (PK)

Number of subjects 57 randomized to complete 42 subjects

Dosing Test or Reference drug (EQ 10mg) base sublingual tablets are to be taken twice daily, once in the morning and once in the evening, for a period of 7 days before crossing-over to receive the next drug assigned for a period of 7 days, followed by a period of 7 days where the third drug assigned will be received.. There will be a total of three 7-day treatment periods during which each subject will receive the test product in one period and the reference product in two other periods.

To ensure optimal absorption, subjects will be instructed to place the tablet under the tongue and allow it to dissolve completely. The tablet will dissolve in saliva. Tablets will not be crushed, chewed, or swallowed

Housing Subjects will be housed in the clinic or hospital for a multiple days in each period during treatment and the collection of pharmacokinetic samples. Housing will be provided for:

* Day 1 and Day 8 or 15 (12-hour confinement)
* Days 6-7
* Days 13-14
* Days 20-21

Investigators may choose to house subjects during the interim days between specified in-patient clinic visits, either in the clinic or at an appropriate off-site facility such as a hotel or motel. Housing offers may be made to each subject population according to the respective Investigator's judgment as to what is best for his/her patients. Such interim housing is not to be considered as study visits, but will be offered at the discretion of the Investigator to all subjects in his/her clinic, at his/her discretion, and simply to improve subject compliance and attempt to reduce variability.

Subjects will be confined for at least 12 hours after initial dosing of either SAPHRIS® (Asenapine) or Asenapine sublingual tablets. Subjects will be required to remain supine for 6 hours following the initial dose. Subjects may get up briefly in order to relieve themselves.

Washout period There will be no washout period

Sampling time points Blood samples will be collected over a dosing interval on day 7, following preliminary sampling on days 5 and 6 to confirm steady-state conditions. The sampling time points are as follows:

* Day 5 (1 sample)
* Day 6 (1 sample)
* Day 7 (15 samples) 0.0(pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0

Dietary Plan Subjects will fast for at least 8 hours prior to and 4 hours after the administration of the morning dose of the test or reference treatment on day 7 of each period (i.e., the days on which blood samples are to be collected to assess the concentration-time curve). All meals on day 7 will be standardized during the study. Water may be allowed, except for 1 hour before and 1 hour after drug administration, when no liquid will be permitted.

Special requirements

* Subjects will remain in the supine position for the first 6 hours after the first dose, even if they were previously on a stable dose of asenapine maleate.
* Subjects will be adequately hydrated. This may be achieved by administering 240 mL of water before the overnight fast, 240 mL of water one hour before dosing, and beginning no sooner than 1 hour after drug administration, 240 mL of water every 2 hours for 6 hours post-dosing. Subjects will not eat or drink for 10 minutes after drug administration.
* Subjects must be adequately informed of possible cardiovascular adverse effects in the consent form.

Safety Parameters

* White blood cell (WBC) counts will be monitored and asenapine maleate sublingual tablet treatment modified, if necessary, in accordance with the leukopenia, neutropenia and agranulocytosis warning in the labeling of the reference listed drug product.
* Subjects requiring modification of asenapine maleate sublingual tablet treatment will be dropped from the study and provided with prompt medical care.
* Blood pressure, heart rate, and body temperature will be monitored during the study and immediate medical care provided for any significant abnormalities.
* Subject medical histories, physical examination and laboratory reports, and all incidents of possible adverse reactions will be reported.

Analyte(s) to measure Asenapine in plasma

Pharmacokinetic parameters

Asenapine AUC0-tau, Cmax, Tmax, Cmin and %Fluctuation will be estimated for each subject and period using WinNonlin version 5.2 or higher. The trough samples collected just prior to the morning dose on Days 5, 6 and 7 in each period will be evaluated to demonstrate that steady-state has been achieved by the final morning dose in each period.

Statistical Analysis

The primary pharmacokinetic parameters (Cmax, AUC0-tau,) and Cmin will be natural log-transformed (ln) prior to statistical analyses. Any ln-transformed parameter where the observed intra-subject CV for the reference product is at least 30% (swr ≥ 0.294) will be evaluated using the scaled average bioequivalence (SABE) method. The GLM procedure of SAS will be used to conduct the SABE analyses, as well as to estimate the intra-subject CV for the reference product. The statistical model for the GLM procedure will contain only a term for Sequence*Site. The linearized Scaled Average Bioequivalence statistic and the upper 95% Confidence Bound on the statistic will be estimated. The ratio of geometric means (T/R) will also be calculated.

Plasma concentrations at each time point, Tmax, %Fluctuation, and any ln-transformed pharmacokinetic parameter where the observed intra-subject CV of the reference product is less than 30% (swr < 0.294), will be evaluated using the average (unscaled) bioequivalence (ABE) approach will be used. The MIXED procedure of SAS will be used in this case with a statistical model that includes terms for Sequence, Site, Sequence*Site, Subject nested within Sequence*Site, Period nested within Site, Treatment, and if necessary, Treatment*Site. A separate statistical analysis will be done to determine if the Treatment*Site term is statistically significant (p<0.05) and needs to be retained in the model. If this term is not significant, it will be dropped from the statistical model for the definitive statistical evaluation. The ratio of geometric means (T/R) and 90% confidence intervals for the ratio, based on least-squares means from the analysis of the log-transformed PK Parameter, will be calculated.

Bioequivalence criteria Bioequivalence will be concluded for those primary parameters evaluated by SABE if:

* The geometric mean Test-to-Reference ratio falls within the range of 0.800 to 1.250.
* The 95% upper confidence bound on the linearized SABE statistic.

Bioequivalence will be concluded for those primary parameters evaluated by ABE if:

The 90% confidence interval on the geometric mean Test-to Reference ratio is contained within the interval 0.800 to 1.250.

Fluctuation for the test product will be evaluated for comparability with the fluctuation of the reference product.

Report format eCTD

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or non-pregnant female subjects aged 18 to 80 years of age
2. For females of child-bearing potential, the subject must be willing to practice a clinically accepted method of birth control
3. Receiving a stable twice daily dose of Asenapine Maleate EQ 10 mg base sublingual tablets for at least 3 months prior to randomization
4. Subjects will be otherwise healthy as determined by the investigator in reference to physical examination, medical history and routine hematologic and biochemical tests
5. Able to obtain written informed consent for the study by the subject or Subject's Legally Acceptable Representative (LAR). If the subject or his/her LAR is unable to read/write, and impartial witness will be present during the entire consenting process who must append his/her signatures to the consent form

Exclusion Criteria:

1. A history of any clinically significant allergic or adverse reactions to asenapine maleate or any comparable or similar product
2. QTc > 450 msec in male subject or QTc > 470 msec in female subjects at screening
3. Heart rate at screening less than 50 bts/min
4. Hypokalemia (defined as serum or plasma potassium less than 3.5 mM or mEq/L) and/or Hypomagnesaemia (defined as serum magnesium less than 0.7 mEq/L) at screening.
5. A history of severe hepatic impairment, drug induced leukopenia/neutropenia, congenital prolongation of the QT interval, cardiac arrhythmias, myocardial infarction or unstable heart disease
6. Concurrent primary psychiatric or neurological diagnosis, including organic mental disorder, severe tardive dyskinesia, or idiopathic Parkinson's disease
7. A total white blood cell count below 4000/mL, or an absolute neutrophil count below 2000/mL
8. A history of granulocytopenia or myeloproliferative disorders (drug-induced or idiopathic)
9. Significant orthostatic hypotension (i.e., a drop in systolic blood pressure of 30 mm Hg or more and/or a drop in diastolic blood pressure of 20 mm Hg or more on standing)
10. Concurrent use of antihypertensive medication or any medication that can predispose to orthostatic hypotension, unless receiving stable dose of those medications for at least 3 months prior to randomization.
11. A medical or surgical condition that might interfere with the absorption, metabolism, or excretion of Asenapine
12. A history of epilepsy or risk for seizures
13. Concurrent use of other drugs known to suppress bone marrow function
14. Expected changes in concomitant medications during the period of study
15. Positive tests for drug or alcohol abuse at screening or baseline
16. A history of alcohol or drug dependence by Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria during the 6-month period immediately prior to study entry
17. Has participated in another clinical research study within 30 days prior to randomization
18. Compliance with outpatient medication schedule not expected
19. History of multiple syncopal episodes
20. Any other clinically significant condition that the investigator thinks puts the subject at risk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Concentration of study medication in the blood at multiple time-points | 17 Time Points (1 on Day 5, 1 on Day 6, 15 on Day 7)
  The primary outcome of this Study is to show bio-equivalence between Asenapine and SAPHRIS. This will be accomplished by measuring the change in concentration of the study medication in the blood at multiple time-points.

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, MD, Principal Investigator — Collaborative Neuroscience Network, LLC; Robert A Riesenberg, MD, Principal Investigator — Atlanta Center for Medical Research; Kurian Abraham, MD, Principal Investigator — New Hope Clinical Research, Inc.; Evagelos Coskinas, MD, Principal Investigator — Clinical Innovations; James S. McDonough, MD, Principal Investigator — Compass Research North, LLC; Gilbert R. Weiner, DO, Principal Investigator — Advanced Pharma CR, LLC; Jim G. Aukstuolis, MD, Principal Investigator — Woodland International Research Group, Inc.
Locations (7):
- United States (7):
  - Woodland International Research Group, Inc., Little Rock, Arkansas
  - Clinical Innovations, Inc, Costa Mesa, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Compass Research North, LLC, Leesburg, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - New Hope Clinical Research, Charlotte, North Carolina